CLINICAL TRIAL: NCT06329817
Title: Incidence of Regurgitation in Patients Undergoing Intubation in Semi-fowler v/s Supine Position in a Tertiary Care Hospital
Brief Title: Incidence of Regurgitation in Patients Undergoing Intubation in Semi-fowler v/s Supine Position
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pak Emirates Military Hospital (Other)
Responsible Party: Principal Investigator, DR.Talha Arshad, Director Head of Army liver transplant unit, Pak Emirates Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: A/28/ER/532/23
Record Dates: First submitted 2024-03-16; First posted 2024-03-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-06

CONDITIONS: Inguinal Hernia Bilateral

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supine position (Experimental)
  Interventions: Procedure: Incidence of regurgitation in two different position.
- Semi- fowler position (Experimental)
  Interventions: Procedure: Incidence of regurgitation in two different position.

INTERVENTIONS:
Procedure: Incidence of regurgitation in two different position. — Preventing aspiration pneumonia in general anaesthesia in two different position supine v/s semi - Fowler

SUMMARY:
One of the most dreaded complication of general anaesthesia is aspiration of gastric contents after induction of general anaesthesia.Many endeavours and measures have been practiced to reduce the incidence of aspiration pneumonia.One such method is to intubate the patient in semi-fowler or supine posture.My study is aimed to find out safe and best position between these two after induction of general anaesthesia to prevent aspiration pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-60 years of age
* Must be able to talk

Exclusion Criteria:

* patients less than 18 years of age or above 60,
* Pregnant women
* Handicapped individuals
* patients with intestinal obstruction

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-16 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Prevention of aspiration pneumonia | 06 months
  To document incidence of regurgitation

CONTACTS AND LOCATIONS:
Overall Officials: IRB PEMH Rwp, Study Director — CPSP
Locations (1):
- PEMH, Rawalpindi, Punjab Province, Pakistan